CLINICAL TRIAL: NCT06028763
Title: Development of Biomedical Technology for the Treatment of Ankle Cartilage Using Injectable Biocomposite Hydrogel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Scientific Center of Traumatology and Orthopedics named after academician N.D. Batpenov (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP19679620
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Ankle Osteoarthritis
Keywords: Cartilage lesions; Osteoarthritis; Mesenchymal stem cells; Ankle arthroscopy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: 40 participants will divide into 2 groups main and control. Main group (n=20): implantation of heparin-conjugated fibrin hydrogel with autologous MSCs and growth factors (TGF-β1 and BMP-4) into the cartilage defect during arthroscopy.
  Control group (n=20): arthroscopic debridement of the joint with microfracturing (traditional method of treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (main) (Experimental): Treatment consists of 2 stages. 1 stage starts with lipoaspiration of subcutaneous adipose tissue from patients. This tissue will then undergo Mesenchymal Stem Cells (MSC) isolation, cultivation and become a biocomposite hydrogel with growth factors. The 2 stage involves ankle joint arthroscopy using the hydrogel for cartilage therapy. To ensure proper hydrogel fixation, we'll clean cartilage remnants, remove fibrous tissue, and create 10mm deep, 2.5mm diameter microperforations. Cartilage donor site prep during arthroscopy will remove non-viable tissue and establish communication with underlying bone marrow. After stopping bleeding, heparin-conjugated fibrin hydrogel with MSCs and growth factors (TGF-β1 and BMP-4) will be implanted using epinephrine-soaked gauze. Hydrogel gels in 3-5 mins. Ankle joint movement tests will confirm successful implantation. Joint stability, articular congruence, and joint condition will be inspected.
  Interventions: Procedure: Injection of biocomposite hydrogel into ankle's cartilage lesion under arthroscopic control
- Group 2 (control) (Active Comparator): Patients from control group will undergo arthroscopic debridement of the joint with microfracturing (traditional method of treatment).
  Interventions: Procedure: Microfracture of ankle's cartilage lesion under arthroscopic control

INTERVENTIONS:
Procedure: Injection of biocomposite hydrogel into ankle's cartilage lesion under arthroscopic control — Surgical treatment involves the use of an injectable biocomposite hydrogel containing autologous mesenchymal stem cells (MSCs), adipose tissue-derived cells, and chondroinductive growth factors (TGF-β1 and BMP-4) under arthroscopic control
  Arms: Group 1 (main)
Procedure: Microfracture of ankle's cartilage lesion under arthroscopic control — Microfracture involves creating tiny perforations in the damaged cartilage, exposing the underlying bone. This encourages the formation of a healing response, where blood and bone marrow cells fill the holes, forming a repair tissue known as fibrocartilage. This newly formed tissue aims to improve joint function and alleviate symptoms associated with cartilage damage. The procedure is performed under arthroscopic guidance, allowing for precise targeting of the lesion while minimizing trauma to the surrounding tissues.
  Arms: Group 2 (control)

SUMMARY:
This study aims to evaluate the effectiveness of heparin-conjugated gel for treating ankle joint cartilage lesions compared to the conventional microfracture method. It involves 40 participants aged 18 to 65 with localized cartilage defects (Outerbridge II-IV) in the ankle's talus bone.

Participants will be divided into two groups: the main group and the control group. The main group will undergo a two-stage process. Initially, adipose tissue will be collected via lipoaspiration from osteoarthritis patients. This tissue will be used to isolate mesenchymal stem cells (MSCs) and extract growth factors, resulting in a biocomposite hydrogel. In the second stage, arthroscopy will be performed to apply the hydrogel for cartilage treatment.

The control group will undergo standard microfracture surgery, a known cartilage repair method.

The study's main objective is to compare heparin-conjugated gel treatment to microfracture in terms of cartilage repair and patient outcomes. A 12-month follow-up will assess short-term and potential mid-term effects.

Data will be analyzed using Microsoft Excel and Statistica 13.0 for descriptive and comprehensive statistical analysis. Quantitative indicators will be assessed using appropriate tests (Mann-Whitney, Wilcoxon T, χ2) to determine significant differences between groups.

The study addresses key questions: Does heparin-conjugated gel offer better cartilage repair, functional improvement, and pain reduction than microfracture? Does the hydrogel approach better preserve joint integrity and slow degeneration? Are there complications with either method? This study combines cellular and surgical components to explore innovative cartilage lesion treatments. Comparing with microfracture and using a thorough follow-up, it aims to enhance cartilage repair techniques and patient outcomes.

DETAILED DESCRIPTION:
Introduction:

This prospective clinical study aims to investigate the effectiveness of heparin-conjugated gel in treating patients with ankle joint cartilage lesions and to compare its outcomes with the traditional method of microfracture. The study aims to provide valuable insights into novel treatment options for cartilage repair.

Study Design and Participants:

The study plans to enroll 40 male and female patients aged 18 to 65 years with localized defects in the articular cartilage of the talus bone (Outerbridge II-IV) within the ankle joint. Participants will be evenly divided into two groups: the main group and the control group, each comprising 20 participants.

Interventions:

Main Group:

In the main group, participants will undergo a comprehensive two-stage treatment approach:

Stage 1 - Biocomposite Hydrogel Preparation:

Subcutaneous adipose tissue will be collected from patients with signs of ankle joint osteoarthritis through lipoaspiration. The extracted tissue will be transferred to the Kazakh National Center of Biotechnology (Astana, Kazakhstan) for the isolation and cultivation of mesenchymal stromal cells (MSCs). A biocomposite hydrogel, containing MSCs and growth factors (TGF-β1 and BMP-4), will be obtained.

Stage 2 - Arthroscopic Cartilage Therapy:

Participants will undergo arthroscopy of the ankle joint. A heparin-conjugated fibrin hydrogel enriched with MSCs and growth factors will be applied to treat cartilage pathology.

Control Group:

The control group will receive the standard microfracture procedure for ankle cartilage lesion under arthroscopic control.

Follow-Up and Safety Assessment:

A 12-month follow-up period will be implemented to assess short-term and potential mid-term effects. Safety assessment of the heparin-conjugated hydrogel will be based on clinical wound healing assessment, local joint changes, and laboratory data (ESR, white blood cell count, C-reactive protein) 5-7 days post-surgery.

Clinical Evaluation:

The therapeutic efficacy of the heparin-conjugated hydrogel will be evaluated using clinical scales and questionnaires, including the American Orthopedic Foot and Ankle Score (AOFAS) and Visual Analogue Scale (VAS) for joint function and quality of life assessment.

Imaging and Rehabilitation:

Prior to surgery, patients will undergo magnetic resonance imaging (MRI) for defect confirmation and dimension assessment using The Magnetic Resonance Observation of Cartage Repair Tissue (MOCART) scale. Postoperative rehabilitation will be tailored individually based on defect characteristics and patient progress. Axial load on the operated limb will be limited for 6 weeks. Gradual weight-bearing will occur from the 6th to the 12th week.

Postoperative Monitoring:

Cartilage condition and joint health will be monitored postoperatively. Hydrogel survival and cartilage defect closure will be observed using MRI at 6 and 12 months.

Data Analysis:

Statistical analysis will use Microsoft Excel and Statistica 13.0. Descriptive statistics methods will calculate means (M) for parametric indicators, medians (Me) and interquartile ranges (Q25-Q75) for non-parametric indicators, and standard deviations (SD). The Mann-Whitney and Wilcoxon T criteria will assess quantitative differences. The χ2 criterion will assess qualitative parameters. Significance will be considered at p<0.05.

Conclusion:

This study's rigorous design aims to contribute to understanding the effectiveness of heparin-conjugated gel for ankle cartilage repair, offering potential improvements over traditional microfracture. Insights gained from this study may lead to enhanced treatment options for patients with cartilage lesions in the ankle joint.

ELIGIBILITY:
Inclusion Criteria:

* patients with a local defect of articular cartilage of the talus bone (Outerbridge II-IV) of the ankle joint;
* an area of no more than 3 cm2 for a single defect or 20 cm2 for multiple defects of the cartilaginous tissue of the talus bone of the ankle joint;
* voluntary consent to participate in the study.

Exclusion Criteria:

* age 18< and >65
* progressive osteoarthritis of the ankle joint in the late stages;
* synovitis of the ankle joint;
* instability of the ankle joint;
* BMI<29.9;
* presence of non-sanitized foci of chronic infection;
* severe mental illnesses (schizophrenia, psycho-organic syndrome);
* hormonal osteopathy;
* hemiparesis on the side of the proposed operation;
* neoplasms of other localizations with or without metastases;
* absence (refusal) of voluntary consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-10-29 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
The American Orthopedic Foot and Ankle Score | 6; 12 months after surgery
  The American Orthopedic Foot and Ankle Score (AOFAS) is a widely used outcome measure designed to assess the functional status and pain levels of patients with foot and ankle disorders. It provides a standardized way to quantify the impact of musculoskeletal conditions on patients' daily lives. The AOFAS score involves a questionnaire that includes various domains related to pain, function, and alignment of the foot and ankle. The scale includes nine items that can be divided into three subscales (pain, function and alignment). Pain consists of one item with a maximal score of 40 points, indicating no pain. Function consists of seven items with a maximal score of 50 points, indicating full function. Alignment consists of one item with a maximal score of 10 points, indicating good alignment. The maximal score is 100 points, indicating no symptoms or impairments.
Visual Analogue Scale | 6; 12 months after surgery
  The Visual Analog Scale (VAS) is a reliable subjective tool used to assess both acute and chronic pain. Individuals express their pain levels by placing a mark on a 10-centimeter line, visually representing a spectrum ranging from "no pain" to "worst pain". Ratings are derived from self-reported symptoms, where individuals use a single handwritten mark on a 10-centimeter line. This line signifies a spectrum between "no pain" at the left end (0 cm) and the utmost level of pain at the right end (10 cm).

SECONDARY OUTCOMES:
Magnetic resonance imaging of ankle | 6; 12 months after surgery
  To confirm the presence of a cartilage tissue defect, determine its localization and preliminary dimensions, and interpret the results according to The Magnetic Resonance Observation of Cartage Repair Tissue (MOCART) scale. The MOCART classification stands out as one of the commonly employed magnetic resonance scores for assessing postoperative cartilage repair tissue. This score, comprising 9 categories and 29 items, yields a comprehensive evaluation, ultimately generating a cartilage repair tissue score ranging from 0 to 100 points. In this scale, 0 points signify the poorest possible score, while 100 points indicate the most favorable score imaginable.
Complete Blood Count | 5 days after surgery
  A Complete Blood Count (CBC) is a comprehensive blood test that evaluates various components of blood, including red blood cells, white blood cells, and platelets. It provides essential information about the health and composition of the blood. In your case, you're particularly interested in assessing the level of erythrocyte sedimentation rate (ESR) and white blood cell count. The ESR measures the rate at which red blood cells settle in a tube of blood and is often used as a marker of inflammation. The white blood cell count measures the number of white blood cells in a given volume of blood and can indicate immune system function and potential infections. By including these specific parameters in the CBC, you aim to gain insights into inflammation levels and immune responses in the body
C-reactive protein | 5 days after surgery
  C-reactive protein (CRP) test plays a crucial role in monitoring the body's response to the surgical procedure. CRP is a protein produced by the liver in response to inflammation. After surgery, the body's immune system reacts to the surgical trauma, causing inflammation at the surgical site. Elevated CRP levels suggest that inflammation is present, which is a normal part of the healing process following surgery. However, extremely high or prolonged CRP levels could indicate excessive or prolonged inflammation, which might raise concerns about potential complications such as infection or poor wound healing.

CONTACTS AND LOCATIONS:
Locations (1):
- Center of National Scientific center Of Traumatology and Orthopedics named after academician N.D. Batpenov, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No